CLINICAL TRIAL: NCT05979701
Title: Use of Simulation Training Versus Theoretical Learning for the Retention of Knowledge and Skills in the Management of Postpartum Hemorrhage: A Multicenter, Comparative Study in Eastern DRCongo.
Brief Title: Simulation for the Retention of Skills in the Management of Obstetric Hemorrhages
Acronym: SimHPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université Evangélique enAfrique (Other)
Collaborators: University Hospital, Angers (Other Government)
Responsible Party: Principal Investigator, Cikwanine Buhendwa Jean Paul, Principal Investigator, Université Evangélique enAfrique
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 001
Record Dates: First submitted 2023-07-29; First posted 2023-08-07 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-06

CONDITIONS: Postpartum Hemorrhage; Simulation Training; Healthcare Providers
Keywords: OSCE
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theoretical education (No Intervention)
- Theoretical education PLUS simulation training (Experimental)
  Interventions: Other: Simulation training

INTERVENTIONS:
Other: Simulation training — The intervention will consist of training participants through simulation in addition to theoretical training. The simulation will cover 3 themes, including diagnosis of haemorrhage, communication between healthcare providers, management of post-partum haemorrhage and transfusion monitoring.
  Arms: Theoretical education PLUS simulation training

SUMMARY:
The aim of this study is to evaluate the retention of knowledge and skills after theory+simulation training versus theoretical training alone in postpartum haemorrhage immediately, 3 months and 6 months after training in South Kivu, in the east of the Democratic Republic of Congo.

ELIGIBILITY:
Inclusion Criteria:

* Work in one of the selected maternity units
* Have two years' experience
* Be either a gynaecologist, obstetrician, general practitioner, midwife, nurse, anaesthetist or laboratory technician.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Score obtained before training and immediatly after training | Before and immediatly after training
  Difference of mean score obtained before training, immediatly after training using validate qestionnaire
Score obtained before training and 3 months after training | 3 months after training
  Difference of mean score obtained before training and 3 months after training using validated questionnaire
Score obtained before training and 6 months after training | 6 months after training
  Difference of mean score obtained before training and 6 months after training using validated questionnaire

SECONDARY OUTCOMES:
OSCE (Objective Structural Clinical Exam) Score | Immediatly and 6 months after training
  Difference of OSCE mean score obtained before training and 6 months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cikwanine JPB, Mukwege D, Mongwa J, Shalamba EM, Maroyi R, Yoyu JT, Martin L. An assessment of the effects of simulation training on management of postpartum hemorrhage: short- and long-term impact on knowledge retention, skills and teamwork in the Democratic Republic of Congo. BMC Med Educ. 2025 May 26;25(1):774. doi: 10.1186/s12909-025-07393-3. PMID 40420075